CLINICAL TRIAL: NCT05747638
Title: Children's Well-being After the COVID-19 Pandemic in French-speaking Primary Schools of the Federation Wallonia - Brussels in Belgium - (DYNAtracs)
Brief Title: Study of Children's Well-being After the COVID-19 Pandemic in Belgian French-speaking Primary Schools
Acronym: DYNAtracs
Status: Active, not recruiting | Type: Observational
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/06DEC/469
Record Dates: First submitted 2023-02-27; First posted 2023-02-28 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Well-being
Keywords: Primary schools
MeSH Terms: interventions — 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Revised Children's Manifest Anxiety Scale (RCMAS) — All participants will be invited to complete a paper questionnaire.
  Other Names: Hospital Anxiety and Depression Scale (HAD)

SUMMARY:
In order to limit the transmission of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), a significant numbers of measures were taken worldwide. It has been shown that the pandemic and its consequences, such as lockdown and isolation, can have a significant long-term impact on the well-being of children.

This study follows the initial DYNAtracs study on SARS-CoV-2 transmission in primary schools. In Belgium, 2488 children and 444 school attenders in 11 primary schools of the Federation Wallonia Brussels are invited. Every participant will be invited to answer a well-being questionnaire. This study aimed to document the children and workers well-being in the primary schools of Belgium after the COVID-19 pandemic. The results of the study should contribute to improved decision making regarding measures for schools and children well-being in the context of current and future pandemics.

The objective of this study is to document the well-being of children and workers after the COVID 19 pandemic in primary schools of the Federation Wallonia-Brussels.

ELIGIBILITY:
Inclusion Criteria:

* All children between the ages of 6 and 12 years and all school attenders from selected primary schools were invited to participate.

Exclusion Criteria:

* Refusal or absence of written informed consent before enrolment

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Sampling procedure for the initial study Eight schools will be chosen by purposive sampling on three criteria: either high or low size of the school, a school within an area with either a high or a low incidence of SARS-CoV-2 on 06/05/2020, the first wave of COVID-19 in Belgium, and a school with either a high or a low socioeconomic level (Belgian 20-point-scale ISE index superior to thirteen or inferior to seven). As direct partners in the project, the ONE ("Office de la naissance et de l'enfance") and the PSE teams ("Promotion de la Santé à l'Ecole") will give a list of schools corresponding to these three criteria.
  In this present study, the investigators will return to the same schools as in the previous DYNAtracs study.
  All participants will be invited to complete a paper questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety symptoms in children | Once
  Anxiety symptoms measured by the "Revised Children's Manifest Anxiety Scale" after the COVID-19 pandemic. A total anxiety score can be calculated by counting 28 items. The minimum score is 0 and the maximum is 28. The higher the score the greater the susceptibility to anxiety.
Anxiety and depression symptoms in school staff. | Once
  Anxiety and depression symptoms measured by the "Hospital Anxiety and Depression" Scale in adults after the COVID-19 pandemic.The person is invited to choose between 4 responses for each question and the score varies between 0 to 3. A total anxiety and depression score can be calculated for a total of 21 points each. The minimum value is 0 and the maximum is 21. A score under or equal 7 was considered with an absence of anxiety and depression; between 8 to 10 corresponds to an anxious or depressive symptoms; and over 11 indicates a definite state of anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: Annie Robert, Pr, Study Director — Université Catholique de Louvain
Locations (1):
- UCLouvain, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study website — http://www.sesa.ucl.ac.be/Dynatracs/

DOCUMENTS (1):
  • Study Protocol (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT05747638/Prot_001.pdf